CLINICAL TRIAL: NCT05336682
Title: Clinical and Radiographic Evaluation of Lesion Sterilization and Tissue Repair Techniques Versus Conventional Pulpectomy in Primary Molars With Inflammed Pulp A Randomized Clinical Trial
Brief Title: Evaluation of Lesion Sterilization and Tissue Repair Techniques Versus Pulpectomy in Primary Molars With Inflammed Pulp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Hamed AbdElHameed Rabea, Assistant lecturer of Pediatric Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis - Irreversible
Keywords: LSTR; Lesion Sterilization and Tissue Repair; pulpectomy; zinc oxide and eugenol; irreversible pulpitis; vital; primary molars
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LSTR with radicular instrumentation. (Experimental)
  Interventions: Procedure: Lesion Sterilization and Tissue Repair with radicular instrumentation
- LSTR with no radicular instrumentation. (Experimental)
  Interventions: Procedure: Lesion Sterilization and Tissue Repair without radicular instrumentation
- Conventional pulpectomy. (Active Comparator)
  Interventions: Procedure: Conventional pulpectomy

INTERVENTIONS:
Procedure: Lesion Sterilization and Tissue Repair with radicular instrumentation — Coronal and accessible radicular pulp tissue are extirpated using rotary files. After proper drying, the paste is placed in the cavity and the canals.
  Arms: LSTR with radicular instrumentation.
Procedure: Lesion Sterilization and Tissue Repair without radicular instrumentation — Only the coronal pulp is removed, the pulpal floor is covered with triple antibiotic paste with propylene glycol mix.
  Arms: LSTR with no radicular instrumentation.
Procedure: Conventional pulpectomy — Pulp tissue extirpation is done. Biomechanical preparation is done using rotary files with frequent irrigation with Chlorhexidine. The canals are dried using sterile absorbent paper points followed by obturation by the paste of ZOE.
  Arms: Conventional pulpectomy.

SUMMARY:
Group I (Experimental group I): Lesion Sterilization and Tissue Repair with radicular instrumentation.

Coronal and accessible radicular pulp tissue are extirpated using rotary files. After proper drying, the paste is placed in the cavity and canals.

Group II (Experimental group II): Lesion Sterilization and Tissue Repair with no radicular instrumentation.

Only the coronal pulp is removed, the pulpal floor is covered with triple antibiotic paste with propylene glycol mix.

Group III (Control group): Conventional pulpectomy. Pulp tissue extirpation is done. Biomechanical preparation is done using rotary files with frequent irrigation with Chlorhexidine. The canals are dried using sterile absorbent paper points followed by obturation by the paste of Zinc oxide and eugenol.

DETAILED DESCRIPTION:
The principal investigator will carry out all treatment procedures, and the patients will be assigned into three groups.

For the three interventions "Two test arms and one control group":

1. Diagnostic chart with personal, medical and dental history will be filled.
2. Clinical examination will be performed to assess the clinical inclusion criteria.
3. Preoperative radiographs will be taken to assess the inclusion criteria. Preoperative radiograph will serve as a reference for the follow-up radiographs.
4. Informed consent is taken from participating parents, and they are asked to attend follow-up meetings every 3 month or whenever there is any symptom.
5. Baseline records (personal data collection, photographs, percussion test and preoperative periapical radiographs).
6. Allocation (concealed by withdrawing a sealed opaque envelope containing eight times folded paper containing the intervention that will be used then writing patient name and I.D. on it and will be opened after performing the access cavity).
7. Administration of Ibuprofen in age-dosage volume before administration of local anesthesia by 30 minutes to decrease pulpal pain, pain of injection and post-operative pain.
8. Administration of local anesthesia at the side of the affected molar.
9. Application of rubber dam for isolation, then a standardized pulpotomy procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation followed by irrigation with 2% Chlorhexidine gluconate. Ethylenediaminetetraacetic acid "EDTA" will be used to remove the smear layer leading to clean and patented dentinal tubules.
10. Children will then be allocated into either one of the groups alternatively depending on the technique of intervention by opening a closed white envelope that is drawn for the patient.

Preparation of triple antibiotic paste:

The commercially available antibiotics are taken in separate dappen dishes. The enteric coating of the tablet is removed by scraping the coating with a blade, and for the capsule the outer capsular material is removed. Then each of the components is powdered separately with a clean mortar and pestle. Care should be taken to avoid wetting of powder. At this stage, the powder can be stored separately in tightly capped containers in a dark place or in the refrigerator to prevent exposure to light and moisture. After proper pulverization, each of the components is taken in a clean glass slab/mixing pad. Then a part of propylene glycol as a solvent is dispensed and mixed with equal parts of antibiotics powder to ensure uniform consistency of the mix. The final preparation will be a soft ball-like structure of 1 mm diameter. Resultant opaque paste has to be stored in airtight containers. If the mix turns translucent on storage, it has to be discarded.

Group I (Experimental group I): LSTR with radicular instrumentation. Coronal and accessible radicular pulp tissue are extirpated using rotary files. After proper drying, the paste is placed in the cavity and canals.

Group II (Experimental group II): LSTR with no radicular instrumentation. Only the coronal pulp is removed, the pulpal floor is covered with triple antibiotic paste with propylene glycol mix.

Group III (Control group): Conventional pulpectomy. Pulp tissue extirpation is done. Biomechanical preparation is done using rotary files with frequent irrigation with Chlorhexidine. The canals are dried using sterile absorbent paper points followed by obturation by the paste of ZOE.

For all groups:

* The molar is then restored with glass ionomer and stainless steel crown.
* Intraoral periapical radiographs are taken after completion of the procedure.
* The children are recalled for clinical evaluation at the interval of 3,6,9,12 months; and radiographic evaluation at 6,12 months.

ELIGIBILITY:
Inclusion Criteria:

* Molars should be restorable.
* Mandibular second primary molars with deep caries, vital carious pulp exposure, irreversible pulpitis.
* Mobility: Non or grade I.
* Radiographic signs of minimal external root resorption.

Exclusion Criteria:

* Children with known allergy to the agents used.
* Children with infective endocarditis.
* Refusal of participation.
* Unable to attend follow-up visits.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Clinical success "binary" | 12 months
  Absence of • Spontaneous pain.
  * Sensitivity to percussion using dental mirror, pain on biting.
  * Swelling.
  * Fistula / Exudate.
  * Mobility.
Radiographic success "binary" | 12 months
  Absence of • Absence of furcation or periapical radiolucency.
  • Absence of change in the extent of internal or external root resorption other than physiologic resorption.

SECONDARY OUTCOMES:
Child cooperation | Immediately after the intervention
  Continuous outcome measured on Frankl's scale immediately after the procedure.
Parental satisfaction | Immediately after the intervention
  Binary outcome measured by direct questioning to parents. "Yes/No"
Chair side time | Immediately after the intervention
  Continuous outcome measured in minutes using stopwatch. (After hemostasis is achieved, time will be measured with a stopwatch from the start of the three techniques till the final restoration is performed)

CONTACTS AND LOCATIONS:
Overall Officials: Gihan M Abuelniel, Professor, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No